CLINICAL TRIAL: NCT00920335
Title: Adult Intracranial Ependydomas : Prognostic and Diagnostic Factors Assessment and Molecular Characterization
Brief Title: Adult Intracranial Ependymoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-25; 2008-A01289-46
Record Dates: First submitted 2009-05-04; First posted 2009-06-15 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Intracranial Ependymoma
Keywords: Adult intracranial ependymoma
MeSH Terms: conditions — Familial ependymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: tumoral sample — Ependymoma tumoral sample

SUMMARY:
Adult intracranial ependymoma is a relatively rare brain tumour entity, accounting for 2-5% of all intracranial neoplasms. The pertinent prognostic factors as well as the pattern of recurrence remain to be elucidated. According to several recent reports, the prognostic value of Karnofski performance status, tumour location, the extent of surgical removal, histological grade and even postoperative radiotherapy remain controversial. As a consequence, optimal therapeutic management of adult intracranial ependymomas remains an ongoing debate. For this reason, a retrospective study conducted by the French society of neurosurgery (SFNC), neuropathology (SFNP) and the association of the neuro-oncologists of French expression (ANOCEF) was undertaken and allowed to collect 258 cases coming from 25 centers, initially diagnosed as intracranial ependymomas between 1990 and 2004. Clinical and follow-up data of these patients are known and the paraffin embedded samples as well as the frozen tissues available have been centralized. Central pathological review of these 258 cases was conducted by two senior neuropathologists and confirmed the diagnosis of ependymoma in 152 cases, thus constituting the most important series of the literature. Few molecular studies were carried out on ependymomas. The investigators have the opportunity, based on this important series, to determine the clinicopathological criteria and the molecular markers who will allow a better characterization of the diagnosis and the prognosis of these tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis later(posterior) than January, 1990
* Diagnosis previous to June, 2004
* Available postoperative MRI at the not dead patients during operating
* Diagnosis of EICA held(retained) after centralized second reading
* Absence of histories of radiotherapy and\or chemotherapy for a brain damage

Exclusion Criteria:

* Diagnosis previous to January, 1990
* Diagnosis later(posterior) than June, 2004 ·
* Diagnosis of EICA not held(retained) after centralized second reading
* Histories of radiotherapy and\or chemotherapy for a brain damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to identify a gene expression pattern associated with recurrence in adult intracranial ependymomas. | 3 years

SECONDARY OUTCOMES:
Firstly to identify reliable molecular markers of the diagnosis of adult intracranial ependymomas and, secondly, to seek a molecular signature selectively expressed in sub-groups of ependymomas according to topography, age and histological grading. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: philippe METELLUS, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France